CLINICAL TRIAL: NCT05468632
Title: A Multicentre, Single-arm, Retrospective Study Investigating Glycaemic Control in GLP-1 Naive Participants With Type 2 Diabetes Who Initiated Once-weekly Semaglutide (OZEMPIC) in a Real World Setting in North Macedonia
Brief Title: A Study in North Macedonia Investigating Retrospective Data of Glucagon-like Peptide-1 (GLP-1) Participants With Type 2 Diabetes (T2D) in Real World Environment (RWE) Setting (MIRAGE)
Acronym: MIRAGE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9535-4976; U1111-1273-4429 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glucagon like peptide-1 (GLP-1) naive participants with Type 2 Diabetes (T2D): Glucagon like peptide-1 (GLP-1) naive adult type 2 diabetes (T2D) participants who initiated once weekly (OW) semaglutide were treated according to current clinical practice, applicable local labels, and standard of care as per physicians' discretion.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants who initiated once weekly (OW) semaglutide in routine clinical practice in were enrolled in the study. The participants were treated according to current clinical practice, applicable local labels, and standard of care as per physicians' discretion.

SUMMARY:
The purpose of this study is to investigate glycaemic control and other clinical parameters in glucagon like peptide -1 (GLP-1) naive adult participants with type 2 diabetes (T2D) who initiated once weekly (OW) semaglutide in local clinical practice in North Macedonia. The participants were treated according to current clinical practice, applicable local labels, and standard of care as per physicians' discretion. The total duration of the study is planned to be approximately 30 weeks which is the period from OW semaglutide initiation to end of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age above or equal to 18 years at the time of once weekly (OW) semaglutide initiation.
* The decision to initiate treatment with commercially available OW semaglutide has been made by the participant and the treating physician before and independently from the decision to include the participant in this study.
* Adult participants with type 2 diabetes (T2D) initiated with OW semaglutide at least 30 +- 4 weeks prior to data collection.
* Participants should have baseline glycated haemoglobin (HbA1c) measurement and at least one HbA1c measurement after baseline. For baseline HbA1c measurement, the most recent value less than 12 weeks prior to OW semaglutide initiation will be used.

Exclusion Criteria:

* Previous participation in this study.
* Prior use of GLP-1 within last one year.
* Participants with type-1 diabetes and gestational diabetes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Glucagon like peptide-1 (GLP-1) naive adult type 2 diabetes (T2D) participants who initiated once weekly (OW) semaglutide were treated according to current clinical practice, applicable local labels, and standard of care as per physicians' discretion.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of follow-up (week 30+- 4 weeks)
  Measured as percentage (%) point.

SECONDARY OUTCOMES:
Change in body weight | From baseline (week 0) to end of follow-up (week 30+- 4 weeks)
  Measured in kilograms (kg).
Change in body weight | From baseline (week 0) to end of follow-up (week 30+- 4 weeks)
  Measured as percentage (%).
Change in waist circumference | From baseline (week 0) to end of follow-up (week 30+- 4 weeks)
  Measured in centimeter (cm).
Change in fasting plasma glucose (FPG) | From baseline (week 0) to end of follow-up (week 30+- 4 weeks)
  Measured in millimoles per liter (mmol/l).
Change in Lipid parameters (total cholesterol, low density lipoprotein cholesterol [LDLc], high density lipoprotein cholesterol [HDLc], triglycerides) | From baseline (week 0) to end of follow-up (week 30+- 4 weeks)
  Measured in millimoles per liter (mmol/L).
Change in Blood Pressure (systolic and diastolic) | From baseline (week 0) to end of follow-up (week 30+- 4 weeks)
  Measured in millimiters of mercury (mmHg).
Glycated haemoglobin (HbA1c) less than 7% | At end of follow-up (week 30 +- 4 weeks)
  Measured as Yes/No.
Reduction in glycated haemoglobin (HbA1c) greater than or equal to (>=) 1% | From baseline (week 0) to end of follow-up (week 30+- 4 weeks)
  Measured as Yes/No.
Weight loss >= 5% | From baseline (week 0) to end of follow-up (week 30+- 4 weeks)
  Measured as Yes/No.
Weight loss >= 3% | From baseline (week 0) to end of follow-up (week 30+- 4 weeks)
  Measured as Yes/No.
HbA1c reduction >= 1% and weight loss of >=3% | From baseline (week 0) to end of follow-up (week 30+- 4 weeks)
  Measured as Yes/No.
Having at least 1 severe hypoglycaemic episode | At end of follow-up (week 30 +- 4 weeks)
  Measured as Yes/No.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (15):
- North Macedonia (15):
  - Novo Nordisk Investigational Site, Bitola
  - Novo Nordisk Investigational Site, Debar
  - Novo Nordisk Investigational Site, General Hospital Kavadarci
  - Novo Nordisk Investigational Site, Gostivar
  - Novo Nordisk Investigational Site, Kičevo
  - Novo Nordisk Investigational Site, Kočani
  - Novo Nordisk Investigational Site, Kumanovo
  - Novo Nordisk Investigational Site, Ohrid
  - Novo Nordisk Investigational Site, Prilep
  - Novo Nordisk Investigational Site, Shtip
  - Novo Nordisk Investigational Site, Skopje
  - Novo Nordisk Investigational Site, Struga
  - Novo Nordisk Investigational Site, Stumica
  - Novo Nordisk Investigational Site, Tetovo
  - Novo Nordisk Investigational Site, Veles

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com